CLINICAL TRIAL: NCT06259006
Title: TREAT-SC: A Randomised, Double-Blinded, Placebo-Controlled Trial of Early, Short Course Oral Dexamethasone for the Treatment of Sydenham Chorea in Children
Brief Title: TREAT-SC: Early, Short Course Oral Dexamethasone for the Treatment of Sydenham Chorea in Children
Acronym: TREAT-SC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Starship Child Health, Te Toka Tumai Auckland (Other Government)
Collaborators: Health Research Council, New Zealand (Other); Menzies School of Health Research (Other)
Responsible Party: Principal Investigator, Hannah F Jones, MD, Paediatric Neurologist, Principal Investigator, Starship Child Health, Te Toka Tumai Auckland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StarshipChild
Record Dates: First submitted 2024-01-22; First posted 2024-02-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Rheumatic Fever; Sydenham Chorea
Keywords: Sydenham Chorea
MeSH Terms: conditions — Rheumatic Fever; Chorea | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Participants will be randomised and allocated 1:1 to blinded dexamethasone or placebo groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be achieved by over-encapsulation of tablets so that placebo cannot be distinguished from dexamethasone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone (Experimental): Participants will receive oral dexamethasone 20mg/m2/day in three divided doses, (maximum dose 24mg/day), for 3 days
  Interventions: Drug: Dexamethasone Oral
- Placebo control (Placebo Comparator): Participants will receive oral placebo tablet three times a day for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone Oral — Dexamethasone suspension (1mg/ml) 20mg/m2/day (maximum dose 24mg/day) given in three divided doses
  Arms: Dexamethasone
Drug: Placebo — Matching capsules taken orally three times daily for three days
  Arms: Placebo control

SUMMARY:
The purpose of this study is to find out whether an early three-day course of an oral steroid medication (dexamethasone) can improve the physical and mental recovery and wellbeing for children with Sydenham's chorea.

Sydenham's chorea is a condition that impacts approximately 12% of children with acute rheumatic fever. It is caused by inflammation in the brain following an abnormal immune response to Group A streptococcus bacterial infection. Sydenham's chorea is a movement disorder that causes children's faces, hands, and feet to move quickly and uncontrollably, and can also affect mood and concentration. The physical recovery from Sydenham's chorea can take two to six months but the mental recovery (e.g. mood and concentration) can take longer to resolve. Sydenham's chorea remains endemic in Māori, Pacific Islander, Aboriginal and Torres Strait Islander children in New Zealand and Australia.

There is limited evidence to direct treatment of Sydenham's chorea, and clinical practice differs widely around the world. Dexamethasone is an oral steroid which targets the abnormal immune response and successfully treats other immune-mediated brain disorders, with good tolerability.

TREAT-SC is a randomized, double-blinded, placebo-controlled trial which will investigate whether a three day course of oral dexamethasone safely and effectively treats the movement disorder and psychiatric symptoms of Sydenham's chorea. The trial will recruit 80 participants from study sites in Australia and New Zealand.

DETAILED DESCRIPTION:
Aim: The aim of the trial is to determine whether an early, short course of oral dexamethasone is a safe and effective treatment to reduce morbidity associated with Sydenham's chorea in New Zealand and Australian children.

Objectives:

* The primary objective is to determine whether oral dexamethasone is an effective treatment to reduce Sydenham's chorea severity in New Zealand and Australian children at one month
* The secondary objectives are to determine whether oral dexamethasone is an effective treatment to reduce Sydenham's chorea severity at different time points, relapse and recurrence rates at three and 12 months, total hospital length of stay at three months, treatment failure at 14 days, use of adjunctive chorea treatments, Universidade Federal de Minas Gerais (UFMG) Sydenham's Chorea Rating Scale (USCRS) subscores, and psychiatric symptoms scored by the Strengths and Difficulties Questionnaire at one, three and 12 months. The safety of oral dexamethasone use will be assessed at study visits on days three and seven and at one month to monitor for any adverse events which may relate to dexamethasone use.

Research Design: TREAT-SC is a pragmatic parallel-group, double-blinded, placebo-controlled, 1:1 randomized efficacy trial comparing a three-day course of oral dexamethasone with placebo to treat Sydenham's chorea in New Zealand and Australian children. TREAT-SC will be a multi-site trial with participants recruited from hospitals in New Zealand and Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Sydenham's chorea of any severity diagnosed by a paediatrician or neurologist based on national ARF guidelines
2. Child or adolescents aged 4 years to <18 years of age

Exclusion Criteria:

1. Administered steroids or intravenous immunoglobulin since onset of the current Sydenham's chorea episode
2. Evidence of concomitant severe, acute infection
3. History of hypersensitivity to dexamethasone or its excipients
4. Pregnancy
5. Confirmed exposure of an unimmunised child to measles, mumps, rubella or chickenpox within the previous four weeks
6. Receipt of a live vaccine within the previous four weeks
7. Medical condition or treatment with medication which in the opinion of the trial investigators would make the child unsuitable for the trial

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Chorea severity at 1 month | 1 month
  Chorea severity measured using the Universidade Federal de Minas Gerais Sydenham's Chorea Rating Scale. Scores range from 0 to 108. A higher score correlates with a worse outcome.

SECONDARY OUTCOMES:
Chorea severity | 7 days, 3 months, 12 months
  Chorea severity measured using the Universidade Federal de Minas Gerais Sydenham's Chorea Rating Scale. Scores range from 0 to 108. A higher score correlates with a worse outcome.
Total hospital length of stay | 3 months
  Total hospital length of stay for chorea at three months
Treatment failure at 14 days | 14 days
  Number of participants with treatment failure at 14 days
Use of adjunctive chorea treatments | 1 month
  Number of participants treated with adjunctive chorea treatments
Chorea relapse and recurrence | 3 and 12 months
  Number of participants with chorea relapse and recurrence at 3 and 12 months
Universidade Federal de Minas Gerais Sydenham's Chorea Rating Scale Subscores. | 7 days, 1 month, 3 months, 12 months
  Behaviour (0 to 24 points), Activities of Daily Living (0 to 28 points) and Motor Assessment (0-56 points). A higher score correlates with a worse outcome.
Psychiatric symptoms | 1 month, 3 months and 12 months
  Strength and Difficulties Questionnaire Total Difficulties Score. The resultant score ranges from 0 to 40. An abnormally high total difficulties score correlates with worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah F Jones, MBChB PhD, Principal Investigator — Starship Child Health, Te Whatu Ora Health New Zealand; Kathryn V Roberts, MBBS PhD, Principal Investigator — Royal Darwin Hospital
Locations (17):
- Royal Darwin Hospital, Darwin, Northern Territories, Australia
- New Zealand (16):
  - KidzFirst Hospital, Auckland
  - Starship Child Health, Te Toka Tumai, Auckland, Auckland
  - Waitākere Hospital, Auckland
  - Gisborne Hospital, Gisborne
  - Waikato Hospital, Hamilton
  - Hawkes Bay Fallen Soldiers' Memorial Hospital, Hastings
  - Hutt Hospital, Lower Hutt
  - Wairarapa Hospital, Masterton
  - Taranaki Base Hospital, New Plymouth
  - Palmerston North Hospital, Palmerston North
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital, Wellington
  - Whakatāne Hospital, Whakatāne
  - Whanganui Hospital, Whanganui
  - Whangārei Hospital, Whangarei

IPD SHARING:
Plan to Share IPD: No
De-identified data would be shared with researchers conducting meta-analysis study if robust research plan is provided and request emailed to PI.